CLINICAL TRIAL: NCT01232933
Title: Use of the VasoNova VPS System During PICC Placement in an Algorithm Confirmation Study Using Fluoroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VasoNova, Inc. (Industry)
Responsible Party: Kim Tompkins, VP Regulatory and Clinical Research, VasoNova, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TP-0120
Record Dates: First submitted 2010-06-15; First posted 2010-11-02 (Estimated); Last update posted 2010-11-02 (Estimated); Status verified 2010-11

CONDITIONS: Any Condition Requiring a PICC Placement
Keywords: PICC

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- VPS System (Experimental): Use of navigational VPS system to place catheter
  Interventions: Device: VPS System

INTERVENTIONS:
Device: VPS System — Use of the navigational VPS system during catheter placement

SUMMARY:
Subjects meeting study requirements will be consented and have their PICC catheter placed using navigational technology and the tip placement confirmed with radiographic imaging.

ELIGIBILITY:
Inclusion Criteria:

* Adult with a PICC placement order

Exclusion Criteria:

* Pregnant or nursing
* Abnormal ECG
* Anatomic irregularities or history that would prevent proper placement
* Subject does not consent to photography, release of data and x-ray confirmation
* Subject does not understand or is not willing to sign informed consent for the VPS implant procedure and data release

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2010-06; Primary Completion 2010-09 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Performance target: the catheter tip will be located in the lower 1/3 of the SVC or at the cavoatrial junction as evaluated by fluoroscopy with a VPS bullseye at least 90% of the time | participants are followed until catheter tip confirmation via fluoroscopy is completed which is on average one hour from procedure initiation

SECONDARY OUTCOMES:
The VPS will provide a blue bullseye indicator 80-90% of the time | participants are followed until catheter tip confirmation is completed which is on average one hour from the start of the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Georgetown University Hospital, Washington D.C., District of Columbia, United States